CLINICAL TRIAL: NCT07011329
Title: Brain Alterations Detected by Multiplex MR Imaging in Nasopharyngeal Carcinoma Patients After Treatment
Brief Title: Brain Alterations Based on Multiplex MR Imaging in Nasopharyngeal Carcinoma Patients After Treatment, and Their Correlation With Clinical Cognitive Scores.
Acronym: NPC
Status: Active, not recruiting | Type: Observational
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, Dan Liu, physician-in-charge, Hubei Cancer Hospital
Other Study IDs: LLHBCH2023YN-019
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
Keywords: npc; MTP; Cognitive decline
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Niemann-Pick Disease, Type A; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- before(pre-) and after (post-) treatment groups: The pre-treatment group refers to before treatment, while the post-treatment group refers to after treatment.
  Interventions: Radiation: Changes in the brain MTP parameters after radiotherapy

INTERVENTIONS:
Radiation: Changes in the brain MTP parameters after radiotherapy — Our study explores the changes in brain MTP parameters and their correlation with clinical cognitive scores before and after chemotherapy and/or radiotherapy in patients with NPC. We investigates MRI-derived multiparametric imaging biomarkers (MTP) as predictive biomarkers for chemotherapy/radiotherapy-induced cognitive decline in nasopharyngeal carcinoma, aiming to optimize neurotoxicity risk stratification and guide personalized neuroprotective interventions in precision oncology.

SUMMARY:
The objective of this study is to examine the potential impact of the treatment before, during, and/or after radiotherapy on the brain in patients with nasopharyngeal carcinoma (NPC) using Multiplex (MTP) MR imaging sequence, which generate multiple contrasts with one-time scan. We aimed to investigate the altered MTP parameters and their correlation with clinical cognitive scores before and after the treatment.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is one of the most common malignancies in the head and neck region. Radiotherapy is the primary treatment for NPC patients, particularly those with T3 and T4 stages. However, radiotherapy often induces brain changes during the acute phase, early delayed phase, or late delayed phase, which may even lead to temporal lobe brain injury and subsequent cognitive impairment. Conventional magnetic resonance imaging (MRI) typically fails to detect corresponding radiological alterations in the brain regions affected by these delayed reactions, even when cognitive dysfunction manifests in patients as early as 6 months post-radiotherapy, so as the other treatment. Previous structural MRI studies (e.g., diffusion tensor imaging [DTI], voxel-based morphometry [VBM]) and resting-state functional MRI analyses (e.g., regional homogeneity [ReHo], functional connectivity [FC], graph theory-based methods) have demonstrated that subtle structural changes and functional abnormalities can be observed prior to apparent radiological changes in NPC patients post-radiotherapy. Additionally, radiomics models based on machine learning have shown promise in predicting early radiation-induced brain injury. However, conventional MRI sequences provide limited imaging information, involve cumbersome and complex data processing, and cannot simultaneously integrate multiple imaging modalities or analyze diverse parameters in a single scan. Therefore, developing a novel MRI imaging technique capable of rapidly, simply, and efficiently detecting induction/radiation-induced brain injury or necrosis in NPC patients during the early stages remains a critical challenge for improving survival outcomes and prognosis in clinical practice.

Multiparametric quantitative magnetic resonance imaging (MulTipLex, MTP) is an emerging technique that enables simultaneous acquisition of multiple contrast mechanisms and quantitative physicochemical parameters in a single scan. This technology has been widely applied in the diagnosis and quantitative analysis of neurological disorders such as Alzheimer's disease, Parkinson's disease, temporal lobe epilepsy, and tuberous sclerosis. It has also been utilized for prognostic prediction of cerebral infarction and integrated with multimodal imaging (e.g., PET-MRI, nuclear medicine) to assist in the staging of nasopharyngeal carcinoma, prostate cancer, and cervical cancer. Notably, MTP offers rapid imaging acquisition, mature technical workflows for brain segmentation and quantitative analysis, and comprehensive data fusion capabilities. To date, no studies have investigated the application of MTP in evaluating induction/radiation-induced cognitive dysfunction following NPC before, during, and/or after radiotherapy.

All patients underwent MTP imaging and Montreal Cognitive Assessment (MoCA) tests between different treatment courses.All MRI data were acquired using a 3.0 T MRI scanner (uMRI 790; United Imaging Healthcare, Shanghai, China) equipped with a 32-channel phased-array head coil. A single MTP scan allowing for the acquisition of multiple contrasts, including aT1W, SWI, cPDW, cT1w, T2Star, T1Map, PDMap, R2Star, and quantitative susceptibility mapping (QSM), was collected for each subjec.The MTP data were analyzed using BrainTool software. Then a single-group paired t-test, Pearson's correlations,a two-sample t-test, Receiver operating characteristic curve (ROC) analyses were utilized to analyse those MTP data and clinical data.

We hypothesis the MTP MR sequence can effectively evaluate brain alterations and cognitive impairment in NPC patients following their teratment.

ELIGIBILITY:
Inclusion Criteria:

* pathological evidence of NPC (stages III-IV at diagnosis according to the 8th edition of the UICC/AJCC staging system for NPC)
* right-handed
* prepared to receive treatments
* prepared to receive the Montreal Cognitive Assessment (MoCA)

Exclusion Criteria:

* brain invasion
* brain tumor or atrophy, neural-associated diseases, a history of brain surgery
* any current medications that may affect cognitive function
* inability to attend MRI scanning

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
volume | 3 months
  the brain volume changes after treatment in NPC patients

CONTACTS AND LOCATIONS:
Overall Officials: Zilong Yuan, MD, Study Director — Hubei Cancer Hospital, Tongji Medical College, Huazhong University of Science and Technology; Dan Liu, MD, Study Chair — Hubei Cancer Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Radiology, Hubei Cancer Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
The raw/processed data required to reproduce these findings cannot be shared at this time as the data also forms part of an ongoing study.

REFERENCES:
- See also: United Imaging Healthcare Official Website of uAiFI Techology including brain analysis based on MTP — https://www.united-imaging.com/en/product-service/products/mr
- See also: United Imaging Healthcare Official Chinese Website of uAiFI Techology including brain analysis, which used brainTool software based on MTP — https://www.united-imaging.com/zh-cn/product-service/products/mr